CLINICAL TRIAL: NCT00163306
Title: Complete Remission: Evaluation of the Complete Remission Rates in Patients With Symptomatic Non-erosive Reflux Disease (NERD) or Erosive Gastroesophageal Reflux Disease (GERD) Treated With Pantoprazole 40 Milligram o.d. Over 4 or 8 or 12 Weeks
Brief Title: Efficacy of Pantoprazole in Patients Older Than 18 Years Who Have Symptoms of Acid Reflux (Gastroesophageal Reflux Disease) (BY1023/M3-339)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/M3-339
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Gastroesophageal Reflux Disease; Pantoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
Gastroesophageal reflux disease (GERD) is a medical condition affecting the stomach and esophagus. GERD occurs when the lower esophageal sphincter does not close properly and stomach contents leaks back (refluxes) into the esophagus. GERD is one of the most common medical disorders, with estimates of up to 50% of adults reporting symptoms related to gastric reflux. Proton pump inhibitors (PPI) such as pantoprazole can relieve symptoms of GERD in a large proportion of patients.

When refluxed stomach acidic content touches the lining of the esophagus, it causes a burning sensation in the chest or throat. This sensation is often referred to as heartburn. Some patients have symptoms of GERD without visible destruction of the tissue surface (no visible changes by endoscopic examination).

The aim of the study is to evaluate the effect of pantoprazole on the complete remission of GERD. Complete remission is defined as endoscopically confirmed healing and symptom relief after a maximum of 12-week treatment period. Pantoprazole will be administered once daily in the morning. Endoscopy will be performed at the start of the study, and then as required after 4, 8, or 12 weeks. The study will provide further data on safety and tolerability of pantoprazole.

ELIGIBILITY:
Main Inclusion Criteria:

* Outpatients
* Reflux disease-related symptoms for at least 12 weeks, which need not be consecutive, in the previous 12 months or endoscopically confirmed reflux esophagitis grade A to D, according to LA-classification

Main Exclusion Criteria:

* Regular intake of systemic glucocorticosteroids, NSAIDs including COX-2 inhibitors on >3 consecutive days per week within the previous 28 days; exception: regular intake of acetylsalicylic acid up to a daily dose of 150 mg/day
* Intake of PPIs (proton pump inhibitor) during the last 10 days, of histamine 2-receptor antagonists or prokinetics during the last 5 days, intake of sucralfate during the last 2 days before the start of the study
* Intake of PPIs in combination with antibiotics for eradication of H. pylori during the last 28 days prior to study start
* Eradication of H. pylori during the last 28 days prior to study start
* Acute peptic ulcer and/or ulcer complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2005-05

PRIMARY OUTCOMES:
complete reflux disease remission rate after 8 weeks of treatment defined as symptom relief assessed by reflux questionnaire (ReQuest Trademark) and endoscopically confirmed healing.

SECONDARY OUTCOMES:
complete reflux disease remission rates after 4, 8, and 12 weeks
time to reach first complete remission
time to reach sustained complete remission
time to reach first symptom relief that is based on the pre-defined GERD symptoms threshold of the reflux questionnaire
average symptom load above pre-defined GERD symptoms threshold
relief rates from reflux disease related complaints after 4, 8 and 12 weeks
endoscopically confirmed healing rates after 4, 8, and 12 weeks
symptom relief rates after 4, 8 and 12 weeks
influence of the H. pylori status on the complete reflux disease remission rate
influence of the H. pylori status on the symptom relief rates
influence of the H. pylori status on the endoscopically confirmed healing rates.

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Heinze, MD, Study Chair — Altana Pharma AG, D-78467 Konstanz, Germany, info.clintrials@altanapharma.com
Locations (68):
- Austria (8):
  - Altana Pharma/Nycomed, Deutschlandsberg
  - Altana Pharma/Nycomed, Feldbach
  - Altana Pharma/Nycomed, Graz
  - Altana Pharma/Nycomed, Krems A. D. Donau
  - Altana Pharma/Nycomed, Lilienfeld
  - Altana Pharma/Nycomed, Stockerau
  - Altana Pharma/Nycomed, Vienna
  - Altana Pharma/Nycomed, Wiener Neustadt
- Germany (37):
  - Altana Pharma/Nycomed, Amberg
  - Altana Pharma/Nycomed, Aschersleben
  - Altana Pharma/Nycomed, Bad Bramstedt
  - Altana Pharma/Nycomed, Bad Schwalbach
  - Altana Pharma/Nycomed, Beckum
  - Altana Pharma/Nycomed, Berlin
  - Altana Pharma/Nycomed, Flensburg
  - Altana Pharma/Nycomed, Freiburg im Breisgau
  - Altana Pharma/Nycomed, Freising
  - Altana Pharma/Nycomed, Germersheim
  - Altana Pharma/Nycomed, Hamburg
  - Altana Pharma/Nycomed, Haßfurt
  - Altana Pharma/Nycomed, Herzogenrath
  - Altana Pharma/Nycomed, Jülich
  - Altana Pharma/Nycomed, Kirchheimbolanden
  - Altana Pharma/Nycomed, Landsberg
  - Altana Pharma/Nycomed, Langen
  - Altana Pharma/Nycomed, Leipzig
  - Altana Pharma/Nycomed, Ludwigsburg
  - Altana Pharma/Nycomed, Ludwigshafen
  - Altana Pharma/Nycomed, Lübeck
  - Altana Pharma/Nycomed, Lütjenburg
  - Altana Pharma/Nycomed, Magdeburg
  - Altana Pharma/Nycomed, Mönchengladbach
  - Altana Pharma/Nycomed, München
  - Altana Pharma/Nycomed, Nieder-Olm
  - Altana Pharma/Nycomed, Oelde
  - Altana Pharma/Nycomed, Potsdam-Babelsberg
  - Altana Pharma/Nycomed, Reinfeld
  - Altana Pharma/Nycomed, Rottweil
  - Altana Pharma/Nycomed, Saarbrücken
  - Altana Pharma/Nycomed, Schweinfurt
  - Altana Pharma/Nycomed, Stuttgart
  - Altana Pharma/Nycomed, Tessin
  - Altana Pharma/Nycomed, Wiesbaden
  - Altana Pharma/Nycomed, Wolfsburg
  - Altana Pharma/Nycomed, Wolmirstedt
- Hungary (14):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Győr
  - Altana Pharma/Nycomed, Gyula
  - Altana Pharma/Nycomed, Hatvan
  - Altana Pharma/Nycomed, Kaposvár
  - Altana Pharma/Nycomed, Miskolc
  - Altana Pharma/Nycomed, Pécs
  - Altana Pharma/Nycomed, Szeged
  - Altana Pharma/Nycomed, Szekszárd
  - Altana Pharma/Nycomed, Szentes
  - Altana Pharma/Nycomed, Székesfehérvár
  - Altana Pharma/Nycomed, Szombathely
  - Altana Pharma/Nycomed, Tatabánya
  - Altana Pharma/Nycomed, Vác
- Poland (9):
  - Altana Pharma/Nycomed, Bydgoszcz
  - Altana Pharma/Nycomed, Drezdenko
  - Altana Pharma/Nycomed, Kielce
  - Altana Pharma/Nycomed, Krakow
  - Altana Pharma/Nycomed, Rzeszów
  - Altana Pharma/Nycomed, Sopot
  - Altana Pharma/Nycomed, Słupsk
  - Altana Pharma/Nycomed, Torun
  - Altana Pharma/Nycomed, Tychy